CLINICAL TRIAL: NCT06634667
Title: Efficacy and Safety of Third-generation EGFR-TKI Combined With Anlotinib as Maintenance Therapy Following 4-6 Cycles of Chemotherapy and Immunotherapy in NSCLC With Small Cell Transformation After EGFR-TKI Resistance: a Single-arm Prospective Phase II Study
Brief Title: Third-generation EGFR-TKI Plus Anlotinib as Maintenance for NSCLC With Small Cell Transformation After EGFR-TKI Resistance
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20241006
Record Dates: First submitted 2024-10-06; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The experimental cohort (Experimental): third-generation EGFR-TKI combined with anlotinib
  Interventions: Drug: third-generation EGFR-TKI combined with anlotinib

INTERVENTIONS:
Drug: third-generation EGFR-TKI combined with anlotinib — third-generation EGFR-TKI combined with anlotinib as maintenance therapy following 4 to 6 cycles of chemotherapy and immunotherapy until progressive disease.

SUMMARY:
This study aimed to evaluate the efficacy and safety of third-generation EGFR-TKI plus anlotinib as maintenance after chemotherapy plus immunotherapy in advanced NSCLC with small cell transformation after EGFR-TKI resistance.

DETAILED DESCRIPTION:
This prospective interventional clinical study aims to evaluate the efficacy and safety of third-generation EGFR-TKI combined with anlotinib as maintenance therapy following 4-6 cycles of chemotherapy and immunotherapy in patients with advanced NSCLC who developed small cell transformation after EGFR-TKI resistance.Approximately 30 non-small cell lung cancer patients who developed small cell transformation after EGFR-TKI resistance were enrolled and treated with 4-6 cycles of chemotherapy plus immunotherapy followed by maintenance therapy with third-generation EGFR-TKI combined with anlotinib.The study is expected to commence recruitment in mainland China in about November 2024. It is expected that the trial will end in December 2026.

ELIGIBILITY:
Inclusion Criteria:

* 1. Understand the requirements and contents of the clinical trial, and provide a signed and dated informed consent form.
* 2. Age ≥ 18 years.
* 3. Histopathology is confirmed non-small cell lung cancer .
* 4.Patients with advanced non-small cell lung cancer (NSCLC) who experienced small cell transformation after EGFR-TKI resistance.
* 5. Predicted survival ≥ 12 weeks. .
* 6. ECOG 0-2.
* 7. Adequate bone marrow hematopoiesis and organ function.

Exclusion Criteria:

* 1. History of other malignant tumors within 2 years.
* 2. Adverse events (except alopecia of any degree) of CTCAE > grade 1 due to prior treatment (e.g., adjuvant chemotherapy, radiotherapy, etc.) prior to the first dose.
* 3. History of stroke or intracranial hemorrhage within 6 months prior to the first dose.
* 4. The presence of any severe or poorly controlled systemic disease, including poorly controlled hypertension and active bleeding in the judgment of the investigator.
* 5. Subjects with persistent or active infection, including but not limited to hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV) and COVID-19 infection.
* 6. Heart-related diseases or abnormalities
* 7. Past history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy or interstitial lung disease with active clinical symptoms, immune pneumonia caused by immunotherapy.
* 8. Refractory nausea and vomiting, chronic gastrointestinal disease, difficulty swallowing drugs, or inability to adequately absorb sunvozertinib or anlotinib due to previous bowel resection.
* 9. Live vaccine was given 2 weeks before the first medication.
* 10. Women who are breastfeeding or pregnant.
* 11. Hypersensitivity to the test drug and the ingredients.
* 12. Other conditions assessed by the investigator to be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | Time from standard chemotherapy plus immunotherapy to study completion, or up to 36 month
  PFS was defined as the duration from the start of standard chemotherapy plus immunotherapy to disease progression or last follow up

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Time from standard chemotherapy plus immunotherapy to study completion, or up to 36 month
  To assess overall response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as the proportion of subjects who have a complete response (CR) or a partial response (PR)
Adverse events (AEs) according to CTCAE 5.0 | Time from standard chemotherapy plus immunotherapy to study completion, or up to 36 month
  Number of participants with adverse events (AEs) according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Yongchang Zhang, Changsha, Hunan, China